CLINICAL TRIAL: NCT04238351
Title: Effect of Transnasal Humidified Rapid Insufflation Ventilator Exchange During Anesthesia Induction With Double Lumen Endotracheal Tube
Brief Title: Transnasal Humidified Rapid Insufflation System for Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Gil2019-2
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Applying Transnasal humidified rapid insufflation ventilator exchange
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care giver and outcome assessor can not know the group assingment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): usual mask ventilation during anethesia induction
  Interventions: Device: Conventional face mask
- THRIVE (Active Comparator): Applying Transnasal humidified rapid insufflation ventilator exchange during anesthesia induction
  Interventions: Device: Transnasal humidified rapid insufflation ventilator exchange

INTERVENTIONS:
Device: Transnasal humidified rapid insufflation ventilator exchange — applying 40L of oxygen for 1min and afte that increase oxygen flow up to 70L for 1 min.
  Arms: THRIVE
Device: Conventional face mask — applying oxygen using usual face mask
  Arms: Control

SUMMARY:
Transnasal humidified rapid insufflation ventilator exchange (THRIVE) or not during the anesthesia induction

DETAILED DESCRIPTION:
Control group-usual mask ventilation during apnea for anesthetic intubation and check tube positioning THRIVE group-applying THRIVE during apnea for anesthetic intubation and check tube positioning

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled for elective lung surery with one lung ventilation

Exclusion Criteria:

* suspicious difficult intubation (BMI >35kg/m2, mouth opening < 3 finger, Mallampati G >3), Room air SpO2 < 90%, active pulmonary infection, emergency operation, pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-25 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Desaturation | during the anesthesia induciton
  number of patients who experienced SpO2 under 93%

IPD SHARING:
Plan to Share IPD: No